CLINICAL TRIAL: NCT02378090
Title: An Observational Study to Determine the Causes and Identify Increases in Influenza-Like Illness (ILI) in Mexico: The Mexican Emerging Infectious Disease Clinical Research Network (La Red)
Brief Title: A Study to Determine the Causes and Identify Increases in Influenza-Like Illness (ILI) in Mexico
Status: Completed | Type: Observational
Sponsor: Mexican Emerging Infectious Diseases Clinical Research Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: ILI-2014
Record Dates: First submitted 2015-02-16; First posted 2015-03-04 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Influenza Nos or Influenza-like Illness; Acute Respiratory Infections
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will only be identified by the unique identifier assigned to each participant for the study. All repository samples will be stored for a maximum of 15 years after the last enrollment into the study; any remaining samples after this time will be destroyed, following Mexican and United States of America (USA) Federal regulations.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to characterize individuals in Mexico who seek medical care for influenza-like illness (ILI) and Severe Acute Respiratory Infection (SARI), describe seasonal pattern of the pathological agents associated with ILI and SARI and to identify changes in severity of disease caused by a specific agent.

DETAILED DESCRIPTION:
The La Red Network clinical sites will enroll individuals presenting with ILI symptoms. A systematic sample will be chosen across all sites, with the goal of choosing 3 subjects who are outpatients and 3 subjects who are hospitalized every week at each site. It is recognized that, during seasons of low ILI activity, this enrollment goal may not be achieved. To be eligible for selection, subjects must be willing to sign informed consent, or provide informed consent/assent in the case of minors.

Subjects will be followed for a period of 28 days after enrollment to assess vital status. It is estimated that this study will enroll a maximum of 1872 subjects per year for an approximate 7488 subjects in the four years that the study proposes to enroll, depending upon the extent of ILI occurring during the period of this study.

Nasopharyngeal swabs, sputum samples, and blood samples will be obtained at enrollment. The nasopharyngeal swabs and, in adults > 18 years of age, portion of the blood for serum and peripheral blood mononuclear cells (PBMC) will be obtained for storage and shipped to the central repository located at the Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán for respiratory pathogen testing including real-time Polymerase Chain Reaction (PCR) and multiplex techniques.

All enrolled subjects will be assessed at enrollment, at 7 days (+3 days) and at 28 days (+/- 5 days) after enrollment to assess disease resolution and vital status.

The purpose of the study is to provide information regarding the pathogens causing ILI among patients seeking care at the La Red Network sites. The systematic collection of data over time will allow for the determination of seasonal patterns of different etiologic agents and the ability for early identification of the emergence of particular viruses, as well as the ability to identify changes in severity of disease signaled by an increase of severity, hospitalization and/or death attributable to a specific pathogen.

One important aspect of influenza infection is to the need to identify genetic factors associated with severity among patients who present with influenza and develop severe disease. Subjects will be given the option to opt out of the genetic testing by noting it on the informed consent form. This testing will be limited to studies related to respiratory viruses and influenza, and any study designed to use genetic testing. These studies will be submitted for review by the institutional review boards (IRBs) of the sites participating in the La Red Network.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by participant. In pediatric subjects, signed informed consent by the parent(s) or legal guardian(s) and, as required by the Institutional Ethics Committee (IEC), signed assent by participant.
* An acute respiratory infection with:

  * Measured fever of ≥ 38°C or history of fever;
  * Cough; and
  * Onset within the last 10 days.

Exclusion Criteria:

* Onset of ILI illness while hospitalized for any other cause to avoid enrollment of potential nosocomial infections (nosocomial).
* Subjects previously included in this study within the last 30 days of enrollment.
* Having been cared for in the hospital for a period >24 hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected from hospitalized (within the last 24 hours) patients and outpatients that seek medical care due to ILI at the sites of La Red Network and meet inclusion criteria. Those who accept participation will be invited to participate, the study will be explained and informed consent will be obtained. The study population will include children and pregnant women.
Sampling Method: Probability Sample
Enrollment: 888 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Etiologic agents causing ILI and SARI among patients seeking medical care at participating sites in Mexico. | 4 years
  Difference in the proportion of a determined isolated etiologic agent (or hospitalization) in the current 2 weeks (increases) in relation to the prior 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Galindo-Fraga, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Daniel Noyola, MD, Study Chair — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (6):
- Mexico (6):
  - Hospital General y de Alta Especialidad Manuel Gea Gonzalez, Mexico City, D. F.
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, D. F.
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, D. F.
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City, D. F.
  - Instituto Nacional de Pediatria, Mexico City, D. F.
  - Hospital Central Dr. Ignacio Morones Prieto/ Universidad Autonoma de San Luis Potosi, San Luis, Potosi